CLINICAL TRIAL: NCT00163280
Title: Randomised Double-Blind Placebo-Controlled Study of Orally Administered ATL-104 to Assess Safety, Tolerance and Effect on Oral Mucositis in Patients Following Treatment With Chemotherapy and Peripheral Blood Stem Cell Transplant (PBSCT)
Brief Title: Safety, Tolerability and Efficacy of ATL-104 in Oral Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alizyme (Industry)
Responsible Party: Research and Development Director, Alizyme
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ATL-104/034/CL
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-02

CONDITIONS: Mucositis
Keywords: Mucositis; Peripheral blood stem cell transplant
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): ATL-104 50mg
  Interventions: Drug: ATL-104
- 2 (Experimental): ATL-104 100mg
  Interventions: Drug: ATL-104
- 3 (Experimental): ATL-104 150mg
  Interventions: Drug: ATL-104
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: ATL-104

INTERVENTIONS:
Drug: ATL-104 — Daily does of ATL-104 (50,100 or 150mg) or placebo for 3 days prior to the start of chemotherapy and peripheral blood stem cell transplantation. Following stem cell transplantation patients received 3 further daily doses of ATL-104 (50, 100 or 150mg) or placebo.

SUMMARY:
This purpose of this study is to investigate whether ATL-104 is safe and well tolerated, and whether it shows evidence of efficacy in mucositis in patients undergoing PBSCT

DETAILED DESCRIPTION:
Mucositis is a serious side effect of cancer therapy and Peripheral Blood Stem Cell Transplant (PBSCT) which requires appropriate and effective management. Mucositis is a condition in which there is inflammation and ulceration of the mouth, throat and gut caused by damage to the mucosal barrier induced by chemo- and radiotherapy. Symptoms include pain, nausea, abdominal cramping, and vomiting. This study will investigate whether ATL-104, when administered as a swallowable mouthwash, is safe and well tolerated in patients undergoing PBSCT and to investigate its potential to reduce the level of severity of mucositis associated with PBSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haematological malignancies undergoing chemotherapy in association with PBSCT

Exclusion Criteria:

* Clinically significant conditions that would exclude the patient receiving chemotherapy in association with PBSCT
* Visible oral disease
* Significantly reduced platelet and neutrophil count

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse events | 28 days post-treatment
Efficacy: Oral mucositis scale | 28 days post-treatment

SECONDARY OUTCOMES:
Safety: Laboratory monitoring, vital signs, ECG | 28 days post-treatment
Pharmacokinetics of ATL-104

CONTACTS AND LOCATIONS:
Overall Officials: Robert Marcus, Principal Investigator — Addenbrooke's Hospital, Cambridge, UK
Locations (8):
- United Kingdom (8):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Oxford
  - Research Site, Plymouth